CLINICAL TRIAL: NCT06816238
Title: Smart Education for Major Adverse Cardiovascular Events Prevention and Early Detection
Brief Title: Smart Education for MACE Prevention and Early Detection
Acronym: SEED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SEED
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: High-Risk Stroke Population
Keywords: Stroke Prevention; Interactive Education; Medical Knowledge Model; Intelligent Medical Agents; MACE Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): High-risk stroke population receiving interactive education based on a medical knowledge model, utilizing intelligent medical agents and interactive Q&A. The educational content will cover stroke prevention and treatment, tailored to individual risk factors and needs.
  Interventions: Other: Interactive education
- Control Group (Active Comparator): High-risk stroke population receiving traditional health education methods without the use of the interactive medical model and intelligent Q&A system.
  Interventions: Other: Traditional health education

INTERVENTIONS:
Other: Interactive education — interactive education based on a medical knowledge model, utilizing intelligent medical agents and interactive Q&A
  Arms: Intervention Group
Other: Traditional health education — traditional health education methods without the use of the interactive medical model and intelligent Q&A system
  Arms: Control Group

SUMMARY:
With its high incidence, recurrence, disability, and mortality, stroke has become a significant health challenge in society today. However, "stroke can be prevented and treated," and high-risk groups for stroke are the primary beneficiaries of stroke prevention and control measures. Yet, these populations often have low awareness of proper stroke prevention and treatment knowledge. The reasons for this may include limited coverage, lack of accessibility, inadequate relevance, and uneven content quality in traditional health education measures.

To address these issues, innovative intervention strategies are needed to explore more effective health education methods. The occurrence of Major Adverse Cardiovascular Events (MACE), such as stroke, can be reduced by improving the knowledge and practical abilities of high-risk populations regarding scientific stroke prevention and treatment. One such strategy is the use of smartphone-based information software, which can break the constraints of time and space, delivering health education knowledge to a broader audience. To enhance accessibility, key knowledge points can be repeatedly delivered to the target population through one-way push notifications and interactive Q&A, allowing for more engaging and flexible learning. In terms of improving pertinence, it is essential to tailor health education delivery to the individual needs of the educatees, considering factors such as age, education level, and risk factors. Furthermore, the quality of health education content must be authoritative, scientifically accurate, easy to understand, and practically applicable. The content should be based on the latest scientific research and professional medical practice, reviewed by authoritative institutions or experts, and should align with the needs of the educated populations for self-health management. Additionally, human and financial costs should be considered when designing such interventions.

In this study, a large-scale medical model based on a stroke prevention and treatment knowledge base, integrated with an intelligent medical system and interactive Q&A, is employed. This approach ensures content quality while minimizing the need for additional manpower in education and Q&A, making the intervention more cost-effective and scalable for widespread use. The purpose of this study is to explore whether the incidence of MACE in a high-risk stroke population receiving interactive medical model education-based on a stroke prevention and treatment knowledge base-is lower than in a group without such interactive education.

DETAILED DESCRIPTION:
With its high incidence, recurrence, disability and mortality, stroke has become an important health challenge facing the society at present. However, "stroke can be prevented and treated," and high-risk groups of stroke are the main beneficiaries of stroke prevention and control and the intervention targets of "health education" measures. Yet, their awareness of correct stroke prevention and treatment knowledge is low. The reasons may be related to the limited coverage, lack of accessibility, lack of pertinence, and uneven content quality of traditional health education measures.

Therefore, we need to adopt innovative intervention strategies to overcome these constraints and explore effective ways of health education. The occurrence of Major Adverse Cardiovascular Events (MACE), such as stroke, can be reduced by improving the knowledge level and practical ability of scientific stroke prevention and treatment in high-risk populations. In this study, the intervention is based on a large medical model using a medical intelligent agent for interactive Q&A. This approach is designed to enhance popularization, accessibility, pertinence, and content quality.

Popularization: The use of smartphone-based information software can break through the limitations of time and space, conveying health education knowledge to a wider audience.

Accessibility: Key knowledge points can be repeatedly delivered to the target audience through one-way pushes of health education content, complemented by interactive Q&A with intelligent medical agents.

Pertinence: Health education content is personalized based on the individual's age, education level, risk factors, and other personal characteristics, ensuring relevance to each educatee.

Content Quality: The educational content is authoritative, scientifically accurate, easy to understand, and practical, drawing from the latest scientific research and professional medical practices, reviewed by authoritative experts and institutions. The intervention ensures that the educated's needs for self-health management are fully considered.

This model leverages the large medical knowledge base and intelligent medical agents to provide personalized, scalable, and cost-effective education, which eliminates the need for additional manpower in education and Q&A. This approach helps reduce costs while enabling large-scale implementation.

The purpose of this study was to explore whether the incidence of MACE in high-risk stroke populations receiving interactive education based on a medical knowledge model and intelligent Q&A is lower than that in a group without such education.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet the definition of a stroke risk group, including those with hypertension, dyslipidemia, diabetes, atrial fibrillation, valvular heart disease, a history of smoking, significant overweight or obesity, physical inactivity, a family history of stroke, or any combination of 8 or more stroke risk factors.

Individuals with a history of one or more transient ischemic attacks (TIAs) or a previous stroke.

Legal capacity to provide informed consent. Permanent residents of Zhejiang Province with Zhejiang Provincial household registration.

Ownership of a smartphone and access to the Alipay app. Voluntary participation and adherence to the principles of informed consent.

Exclusion Criteria:

Illiteracy or difficulty with reading/communication. Medical personnel. Inability to complete the study questionnaire due to physical or cognitive limitations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87376 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
MACE Incidence | 1 year from enrollment
  The occurrence of major adverse cardiovascular events (MACE), including stroke (ischemic or hemorrhagic), myocardial infarction, heart failure, or cardiovascular death, in participants over the 1-year follow-up period. MACE is a composite outcome that captures the broad range of adverse cardiovascular events.

SECONDARY OUTCOMES:
Stroke Incidence | 1 year from enrollment
  The occurrence of new stroke events (ischemic or hemorrhagic) in participants during the 1-year follow-up period.
Hospitalization Due to Cardiovascular Events | 1 year from enrollment
  The number of hospital admissions related to cardiovascular events, including stroke, myocardial infarction, heart failure, or other significant cardiovascular conditions.
Stroke Prevention and Treatment Knowledge | 1 year from enrollment
  Participants' knowledge of stroke prevention and treatment, assessed via surveys or questionnaires.
Blood Pressure Control | 1 year from enrollment
  Proportion of participants maintaining blood pressure within recommended levels (e.g., <140/90 mmHg) as part of stroke and cardiovascular risk management.
Physical Function and Quality of Life (QoL) | 1 year from enrollment
  Assessment of physical function and overall quality of life, measured using standardized scales like the EQ-5D or the SF-36, to understand the impact of the intervention on the participant's daily living and wellbeing.
Adherence to Stroke Prevention Medications | 1 year from enrollment
  Proportion of participants adhering to prescribed medications (e.g., antihypertensives, antiplatelets) for stroke prevention, measured via self-reports or pharmacy refill data.
Smoking Cessation (for smokers) | 1 year from enrollment
  Proportion of smokers who quit smoking within 3 months of the intervention, as assessed by self-report and/or biochemical validation (e.g., carbon monoxide levels, cotinine levels).
Weight Loss (for overweight participants) | 1 year from enrollment
  Proportion of overweight participants who lose at least 5% of their body weight within 3 months, measured via weight records.
Sense of First Aid for Stroke | 1 year from enrollment
  Improvement in participants' knowledge and confidence in providing first aid in the event of a stroke, measured through a standardized questionnaire or skills assessment.
Thrombolysis Use in Ischemic Stroke | 1 year from enrollment
  Proportion of ischemic stroke patients who receive thrombolysis treatment (IV tPA or intra-arterial therapy) within the recommended time window.

IPD SHARING:
Plan to Share IPD: No